CLINICAL TRIAL: NCT05367661
Title: A Phase 1, Single-Center, Randomized, Placebo-Controlled, Double-Blind, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of CHK-336 in Healthy Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CHK-336 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Chinook Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHK336-01
Record Dates: First submitted 2022-04-05; First posted 2022-05-10 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Healthy Volunteers: Single ascending doses (Experimental): Six dose groups ranging from 15mg to 500mg, under fasting condition.
  Interventions: Drug: CHK336; Drug: Placebo
- Part A: Healthy Volunteer: Single Ascending dose under fed condition (Experimental): 60mg under fed condition.
  Interventions: Drug: CHK336
- Part A: Otherwise Healthy volunteer with Class I or Class II obesity, Single Ascending dose (Experimental): 125mg, under fasting condition.
  Interventions: Drug: CHK336; Drug: Placebo
- Part B: Healthy Volunteers: Multiple Ascending doses (Experimental): 5 dose groups with doses ranging from 30mg to 500mg. Given daily for 14 days, under fasting condition.
  Interventions: Drug: CHK336; Drug: Placebo

INTERVENTIONS:
Drug: CHK336 — Tablet
Drug: Placebo — Tablet
  Arms: Part A: Healthy Volunteers: Single ascending doses; Part A: Otherwise Healthy volunteer with Class I or Class II obesity, Single Ascending dose; Part B: Healthy Volunteers: Multiple Ascending doses

SUMMARY:
This study is designed to assess the safety, tolerability, pharmacokinetics and pharmacodynamic effects of an investigational drug (CHK-336) when administered to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers must meet all the following inclusion criteria to be randomized:

1. Male and female adults18 to 45years old, inclusive, at the time of consent.
2. Body mass index (BMI) between 19 and 32 kg/m2, inclusive, (between 30.0 and < 40.0 kg/m2 for SAD Cohort A8) at screening.
3. Contraception use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. All participants (male or female) who are of childbearing potential must agree to use highly effective contraception during the study. Female participants must continue to use highly effective contraception during the study for 30 days after the last dose of study drug. Female participants should not donate oocytes during this time. Male participants with female partners of childbearing potential must continue to use highly effective contraception during the study and for 90 days after the last dose of study drug. Male participants must agree not to donate sperm during this time. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
4. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at screening and Day -3 as well as a negative urine pregnancy test at Day 1 (predose). WOCBP must agree to undergo a pregnancy test during the study
5. Female participants not of childbearing potential must be either surgically sterile (hysterectomy, bilateral salpingectomy and bilateral oophorectomy) or postmenopausal, defined as no menses for 12 months without an alternative medical cause, with follicle-stimulating hormone (FSH) in the postmenopausal range at screening, based on the central laboratory's ranges.
6. Willing and able to provide informed consent and comply with all study visits and procedures including overnight stays in the clinic
7. Willing and able to comply with a pre-specified diet at least 72 hours prior to dose and throughout the study.
8. Negative urine drug, tobacco, and breath alcohol test result at screening and Day-3.
9. Have not used any nicotine-containing product within 3 months prior to the first study drug administration and who are willing to abstain throughout the study.

Exclusion Criteria:

Healthy volunteers must not meet any of the following exclusion criteria to be randomized

1. Any significant medical history including but not limited to hypertension, diabetes, cardiovascular disease, hemolysis, red blood cell disorders, and/or with clinically significant screening results outside the normal range for laboratory testing, vital signs, medical history, electrocardiograms (ECGs), physical examination as deemed by the investigator. Reticulocytes must be within normal range at screening and prior to dosing. Red blood cell (RBC), hemoglobin, and hematocrit must be within 5% of normal range at screening and prior to dosing.
2. Evidence of chronic kidney disease (CKD) defined by an estimated glomerular filtration rate (eGFR) less than 80 mg/mL/1.73m2 based on the CKD epidemiology collaboration (EPI) equation or the presence of proteinuria at screening and prior to dosing.
3. Have any known malignancy or history of malignancy, except for basal cell skin cancer that has been treated and with no evidence of recurrence for at least 3 months prior to the first study drug administration.
4. History of liver disease, Gilbert's syndrome, or abnormal liver function test (AST, ALT, total bilirubin) above the normal reference range at screening and prior to dosing.
5. Any active infection or acute illness within 30 days prior to the first study drug administration.
6. Major surgery or significant traumatic injury occurring within 28 days prior to first dose of study drug. If major surgery occurred > 28 days prior to first dose of study drug, individual must have recovered adequately from any toxicity and/or complications from the intervention prior to the first dose of study drug.
7. Supine systolic blood pressure <90 or >140 mmHg, supine diastolic blood pressure <50 or >95 mmHg, pulse rate <40 or >100 beats per minute (bpm), or elevated body temperature (>38ºC) at screening and check-in
8. History or presence of a clinically significant ECG abnormalities and QTcF >450 ms for males and >470 ms for females, prior to dosing.
9. Positive serology tests for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus (HCV).
10. Use of any prescription, vaccines, supplements/vitamins, or over-the counter medication (with the exception of oral contraceptives) within 7 days prior to the first study drug administration.
11. Treatment with another investigational product within 30 days prior to the first study drug administration or within the expected washout (~5 half-lives) of the investigational product
12. Prior exposure to CHK-336 (including Part A of this study).
13. History or presence of alcohol abuse or drug use within 30 days prior to the first study drug administration and throughout the study
14. Blood donation or significant blood loss within 60 days prior to the first study drug administration.
15. Pregnancy, intent to become pregnant during the course of the study, or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2022-04-08 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of single ascending doses and multiple ascending doses of CHK-336 in HV | Up to 28 days
  Incidence, nature, and severity of adverse events (AEs), adverse events of special interest (AESI), and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetic measure of Cmax | Up to 17 days
  Maximum observed concentration of CHK -336 in plasma under fasted or fed condition
Pharmacokinetic measure of Tmax | Up to 17 days
  Time to maximum observed concentration of CHK-336 in plasma under fasted or fed condition
Pharmacokinetic measure of AUC (0-∞) | Up to 17 days
  The area under the concentration-time curve from time zero extrapolated to infinity (AUC0-∞) of CHK-336 in plasma under fed or fasted condition
Pharmacokinetic measure of AUC for up to 24 hours (AUC0-24) | up to 17 days
  The area under the concentration-time curve from time zero extrapolated to 24 hours post dose (AUC0-24) in plasma under fed or fasted condition
Pharmacokinetic measure of AUC for up to last measurable time point (AUC0-T) | up to 17 days
  The area under the concentration-time curve from time zero extrapolated to last measurable timepoint (AUC0-T) of CHK-336 in plasma under fed or fasted condition
Pharmacokinetic measure of apparent terminal half-life (t1/2) | up to 17 days
  Apparent terminal half-life (t1/2) of CHK-336 in plasma under fasted or fed condition
Pharmacokinetic measure of exposure accumulation ratios of CHK-336 | up to 17 days
  The exposure accumulation defined as the ratio of last dose to single dose AUC0-24h with once a day dosing
Pharmacokinetic measure of exposure accumulation ratios (Cmax) for CHK-336 | up to 17 days
  The exposure accumulation defined as the ratio of last dose to single dose Cmax with once a day dosing
Pharmacokinetic measure of the amount of CHK-336 excreted in urine | Up to 24 hours
  Measure the amount of CHK-336 excreted in urine under fasted condition

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Cox JH, Boily MO, Caron A, Sheng T, Wu J, Ding J, Gaudreault S, Chong O, Surendradoss J, Gomez R, Lester J, Dumais V, Li X, Gumpena R, Hall MD, Waterson AG, Stott G, Flint AJ, Moore WJ, Lowther WT, Knight J, Percival MD, Tong V, Oballa R, Powell DA, King AJ. Characterization of CHK-336, A First-in-Class, Liver-Targeted, Small-Molecule Lactate Dehydrogenase Inhibitor for Hyperoxaluria Treatment. J Am Soc Nephrol. 2025 Apr 7;36(8):1535-1547. doi: 10.1681/ASN.0000000690. PMID 40193200